CLINICAL TRIAL: NCT06225336
Title: A Phase 1/2, Single-Center, Open-Label, Single-Arm Safety, Tolerability, and Efficacy Study of an Auricle and Wedge Subcutaneous Implant Combination Product (AUR-201) in Patients With Unilateral Microtia
Brief Title: Subcutaneous Implant Combination Product (AUR-201) in Patients With Unilateral Microtia (Australia)
Acronym: AUR-201
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Auregen Biotherapeutics, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUR-201-02
Record Dates: First submitted 2024-01-17; First posted 2024-01-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Microtia
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AUR-201 (Experimental): AUR-201
  Interventions: Combination Product: AUR-201

INTERVENTIONS:
Combination Product: AUR-201 — Auricle and wedge subcutaneous implant consisting of 3-D printed autologous auricular sourced chondrocytes in a biopolymer matrix.

SUMMARY:
AUR-201 is indicated for the treatment of Grade II, III, or IV unilateral microtia in patients 8 to 29 years of age.

DETAILED DESCRIPTION:
AUR-201 is an auricle and wedge subcutaneous implant consisting of 3-D printed autologous auricular sourced chondrocytes in a biopolymer matrix.

ELIGIBILITY:
Inclusion Criteria:

1. Child between 8 and 17 years of age (inclusive) at the time the guardian signs the ICF or adult between 18 and 29 years of age (inclusive) at the time of signing the ICF. Note, the implantations of AUR-201 will initially be staggered based on age and completion of specified DSMB evaluations (see Methodology section);
2. Diagnosed with Grade II, III, or IV congenital unilateral microtia requiring complete auricular reconstruction;
3. Naïve to microtia surgery or have had prior failed microtia surgery not involving the TPF flap;
4. Able and willing to adhere to the post-operative wound care instructions (including, but not limited to, wearing protective devices specified by the PI) and the protocol-specified follow-up schedule;
5. Willing to refrain from non-contact sports and contact sports (e.g., football, soccer, rugby, boxing, karate) for 6 and 12 weeks, respectively, following the first implantation surgery, or longer if deemed necessary for healing by the PI. If the PI opts to implant the AUR-201 wedge at a separate subcutaneous location on Day 0 and then 12 weeks later, implants the wedge in the final location, these periods of refraining from non-contact and contact sports will also apply to the second implantation surgery;
6. PI deems the subject an appropriate candidate for the planned AUR-201 biopsy and implantation procedures (i.e., either the TPF flap technique or the pocket technique) and that the subject meets the following criteria:

   1. Healthy auricular cartilage donor site (e.g., conchal bowl site) on contralateral (non-microtic) ear available for biopsy;
   2. Healthy skin tissue at site of planned microtia repair;
7. Healthy (other than for microtia) as determined by the PI based on medical history, physical examinations, body weight, vital signs, 12-lead electrocardiogram (ECG), and safety laboratory tests at screening/pre-biopsy baseline;
8. Negative test results for human immunodeficiency virus 1 (HIV-1), human immunodeficiency virus 2 (HIV-2), hepatitis B virus (HBV), hepatitis C virus (HCV), Treponema pallidum (i.e., syphilis), and West Nile virus 1 (WNV-1) within seven days prior to the biopsy for harvesting auricular cartilage from the contralateral ear;
9. Able to understand the English language;
10. Subject or guardian able to understand the ICF and give informed consent/assent;
11. Subject or guardian signed the ICFs for both this study (Protocol No. AUR-201-02) and the long-term follow-up (LTFU) study (Protocol No. AUR-201-04);
12. Women of childbearing potential (WCBP) must have a negative serum pregnancy test at screening and a negative urine pregnancy test at the pre-biopsy baseline visit;
13. WCBP must agree to abstain from sex or use an adequate method of contraception* from the time of informed consent through the last study visit at 96 weeks post-implantation;
14. Males must abstain from sex with WCBP or use an adequate method of contraception* from the time of informed consent through the last study visit at 96 weeks post-implantation;

    * Adequate contraceptive methods include those with a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as some double barrier methods (condom with spermicide) in conjunction with use by the partner of an intrauterine device, diaphragm with spermicide, oral contraceptives, birth control patch or vaginal ring, or injectable or implanted contraceptives. Abstinence is acceptable only as true abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

A woman that is postmenopausal (≥2 years since last menstrual period) or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) is not considered a WCBP.

Exclusion Criteria:

1. Any comorbidities likely to affect healing or the ability to adhere to the protocol, including:

   1. Burns, trauma, problematic wound healing, or scarring skin malformations at the planned site of microtia repair or the planned site of biopsy collection for auricular cartilage;
   2. Squamous cell carcinoma, basal cell carcinoma, or melanoma at the planned site of microtia repair or the planned site of biopsy collection for auricular cartilage;
   3. Uncontrolled diabetes or hypertension;
   4. History of diabetes requiring amputation or dialysis;
   5. Serious autoimmune disorder, or ongoing immunocompromised state;
   6. Current or recent history (within four weeks prior to initial screening visit) of a clinically significant bacterial, fungal, or mycobacterial infection;
   7. Current clinically significant viral infection;
   8. History of human transmissible spongiform encephalopathies (TSEs), including Creutzfeldt-Jakob disease;
   9. History of Zika virus infection;
   10. Completed treatment of syphilis within 12 months prior to screening;
   11. Uncontrolled acne vulgaris in the area of the planned AUR-201 implantation site;
   12. History of organ transplant;
   13. Major cardiac, pulmonary, renal, hepatic, metabolic, neurologic, or urologic disorders;
2. Predisposition or history of keloid or hypertrophic scar development;
3. Lifestyle activities likely to affect healing or ability to adhere to the protocol (e.g., active contact sports and protective gear that interferes with wearing post-operative silicone molds and plastic ear cup);
4. Diagnosed with any of the following syndromes or conditions:

   1. Treacher-Collins syndrome;
   2. Nager syndrome;
   3. Goldenhar syndrome or hemifacial microsomia plus an occlusal cant of 20 degrees or greater;
   4. Absence of vertical ramus [as diagnosed on physical exam or computed tomography (CT)];
   5. Absence of zygoma (as diagnosed on physical exam or CT);
   6. Significant orbital asymmetry or micro-ophthalmia (as diagnosed on physical exam or CT);
   7. History of major congenital disorder that could impact wound healing or cell expansion from the biopsy sample;
5. Inadequate renal function as indicated by serum creatinine >1.5 x the upper limit of normal (ULN) and either a >50% decrement of blood flow or anatomic abnormalities on renal scan;
6. Any condition which, in the opinion of the PI, places the subject at unacceptable risk if he/she were to participate in the study;
7. Treatment with an immunosuppressant within 6 months prior to screening;
8. Treatment with a chemotherapeutic within 12 months prior to screening;
9. Treatment with isotretinoin within 12 months prior to screening;
10. Treatment with oral steroids within 1 month prior to screening;
11. Current tobacco or illicit drug use;
12. Participation in another interventional (non-observational) clinical study (other than as a documented placebo subject with no interventions at the planned site of biopsy or implantation) within 6 months prior to screening;
13. Additional planned surgical procedures, including piercings, at the microtia or biopsy sites (i.e., beyond the AUR-201 biopsy and implantation procedures with skin grafts) during the subject's planned participation in this study;
14. Pregnant or breastfeeding (or planning to become pregnant or breastfeed during the study);
15. Presence of an implanted hearing enhancement device if it will interfere with the surgical technique (TPF flap or pocket) planned for AUR-201 implantation;
16. Known hypersensitivity to the biopolymer components used in the manufacture of AUR 201, including gellan gum and sodium alginate;
17. Known hypersensitivity to the components in the AUR-201 transport medium, including Dulbecco's Modified Eagle's Medium (DMEM), L-alanyl-L-glutamine, and 2-[4-(2-hydroxyethyl)piperazin-1-yl]ethanesulfonic acid (HEPES);
18. Known hypersensitivity to amide-containing anesthetics;
19. Known hypersensitivity to povidone iodine.

Ages: 8 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 24 weeks
  To assess the safety and tolerability of AUR-201 in patients with unilateral microtia based on Incidence of Treatment-Emergent Adverse Events from the time of biopsy sample collection of auricular cartilage from the contralateral (non-microtic) ear through 24 weeks post-implantation of AUR-201.
  The severity of AEs will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Appearance/Efficacy of the AUR-201 Implant | 24 weeks
  To assess the efficacy of AUR-201 in patients with unilateral microtia based on improvement in overall appearance at 24 weeks post-implantation compared to pre-implantation baseline as determined by review and rating of photographs on a 5-point Likert scale by a panel of blinded independent experts. (All scores are based on a 5-point Likert scores and are represented as follows: 1 = Poor, 2=Fair, 3=Good, 4= Very Good and 5=Excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Dusseldorp, MD, Principal Investigator — Chris O'Brien Lifehouse
Locations (1):
- Chris O'Brien Lifehouse, Camperdown, Australia